CLINICAL TRIAL: NCT04564131
Title: The Effect of Reflexology Massage Applied to Diabetic Neuropathic Pain on Patients Quality of Life
Brief Title: Reflexology in Diabetic Neuropathic Pain Management
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Istanbul Saglik Bilimleri University (Other)
Responsible Party: Principal Investigator, Nesibe Simsekoglu, Principal Investigator, Istanbul Saglik Bilimleri University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: SY200217B06
Record Dates: First submitted 2020-08-28; First posted 2020-09-25 (Actual); Last update posted 2020-09-25 (Actual); Status verified 2020-09

CONDITIONS: Reflexology; Neuropathic Pain
Keywords: Type 2 Diabetes; Quality of Life; Nursing
MeSH Terms: conditions — Neuralgia; Diabetes Mellitus, Type 2 | interventions — Musculoskeletal Manipulations

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- reflexology practice (Experimental): Blood glucose measurement with a glucometer to be provided by the researcher, blood pressure measurement with a digital blood pressure device, and foot temperature measurement with an infrared thermometer will be made. Turkey podiatry foot care guide will be trained under the guidance of the Society of Endocrinology and Metabolism.
  Experimental group participants will be given 10 sessions of reflexology massage twice a week for 5 weeks. A total of three follow-ups will be performed in the 1st session, the 5th session and the 10th session. In the follow-up sessions; VAS, DN4, LANSS, NePIQol scales will be applied, foot assessment and SWMI test will be applied.
  Interventions: Other: Reflexology
- Control (Experimental): Blood glucose measurement with a glucometer to be provided by the researcher, blood pressure measurement with a digital blood pressure device, and foot temperature measurement with an infrared thermometer will be made. Turkey podiatry foot care guide will be trained under the guidance of the Society of Endocrinology and Metabolism. 1. 3. 5. A total of three follow-ups will be done once in the week. In the follow-up sessions; VAS, DN4, LANSS, NePIQol scales will be applied, foot assessment and SWMI test will be applied.
  Interventions: Other: Control

INTERVENTIONS:
Other: Reflexology — * Hands are washed.
  * The individual is provided to be in a comfortable position to lie down or to be in a semi-sitting position.
  * The toes of the patient are crossed and the patient's feet are placed at our chest level when we sit.
  * Depending on the size of the foot, a slightly moisturizing amount of non-allergenic petroleum jelly is taken, and it is spread to provide slipperiness.
  * Exercises to warm and relax the feet for five minutes.
  * General massage is applied to the whole foot for five minutes.
  * Reflexology massage is applied to the application areas for neuropathic pain.
  * The individual is helped to take a comfortable position.
  * Hands are washed.
  Arms: reflexology practice
Other: Control — No intervention was performed to reduce pain in the control group
  Arms: Control

SUMMARY:
Reflexology massage, applied by applying pressure to any point on the feet, is one of the most popular complementary treatments in the world. Given the negative impact of neuropathic pain on quality of life and the limited effectiveness of traditional medicines, it is important to investigate the effects of various complementary therapies available, including reflexology massage. Therefore, the study was planned as a prospective randomized controlled experimental study with a pre-test and post-test design aiming to investigate the effect of reflexology massage for neuropathic pain on pain intensity and quality of life in diabetic individuals.

DETAILED DESCRIPTION:
Pressure will be applied to the relevant reflex areas of the foot based on the individual's pain area. In order to standardize the application, the procedure will start with the left foot and end with the right foot. Both feet will be massaged using petroleum jelly for 5 minutes of relaxation movements, 5 minutes of general foot massage and 5 minutes of standing and reflex area corresponding to the painful body area. 5 more minutes will be applied to the left foot in order to increase the endorphin secretion and reduce the pain by activating the parasympathetic system. Reflexology massage will be applied for a total of 35 minutes in one session. Each reflexology area will be stimulated 15 times, as less than 10 stimulation to a particular reflexology area does not produce any therapeutic effect and more than 20 stimulations will be excessive. A total of 3 follow-ups will be done throughout the study. In the follow-up sessions; Visual Analogue Scale (VAS), Douleur Neuropathique 4 (DN4), The Leeds Assessment of Neuropathic Symptoms and Signs (LANSS) , Neuropathic Pain Impact on Quality-of-Life questionnaire (NePIQoL) scales will be applied, foot assessment and SWMI test will be applied. The 1st follow-up will be done before any intervention in the 1st session, the 2nd follow-up will be done after the reflexology application in the 5th session, and the 3rd follow-up will be done after the reflexology application at the 10th session . There will be a break of at least one day between two sessions to relax the body and eliminate toxins.

ELIGIBILITY:
Inclusion Criteria:

* Those over the age of 18,
* Literate,
* A diagnosis of neuropathic pain associated with Type 2 diabetes,
* Defined pain of at least 4 severity according to the Visual Analogue Scale (VAS),

Exclusion Criteria:

* A diagnosis of disease causing neuropathy (uremia, malnutrition, liver failure, alcoholism, kidney failure, dialysis treatment, oncology patients, vitamin deficiency),
* have a pacemaker,
* Diabetic foot diagnosis,
* who are pregnant,
* Having vision, hearing, cognitive ability disorders and psychosis, Reflexology massage in the last month,
* Receiving medical treatment with an effect that conceals neuropathic pain symptoms,
* Disc herniation,
* Any infectious skin disease (shingles, fungus, etc.),
* Individuals with open lesions / wounds, scar tissue, fractures, dislocations, amputation, edema, hematoma, thrombophlebitis, inflamed and degenerative joint diseases in the lower extremities will not be included in the sample.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 128 (Estimated)
Dates: Start 2021-04-01 (Estimated); Primary Completion 2021-07-01 (Estimated); Study Completion 2022-04-01 (Estimated)

PRIMARY OUTCOMES:
pain intensity | 5 Months
  According to the Douleur Neuropathique 4 Questions (DN4) questionnaire, neuropathic pain score changes to less than 4 points.
pain intensity | 5 Months
  Change of neuropathic pain score to less than 12 points according to The Leeds Assessment of Neuropathic Symptoms and Signs (LANSS) scale.
life quality | 5 Months
  Change of quality of life score higher than 42 points according to the Neuropathic Pain Impact on Quality-of Life Questionnaire (NePIQoL) scale

CONTACTS AND LOCATIONS:
Overall Officials: Nesibe Simsekoglu, RN, Principal Investigator — Saglik Bilimleri University
Locations (1):
- Saglik Bilimleri University, Istanbul, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Silva NCM, Chaves ECL, Carvalho EC, Carvalho LC, Iunes DH. Effect of Foot Reflexology on Capillary Blood Glucose, Tissue Temperature, and Plantar Pressure of Individuals With Diabetes Mellitus (Type 2): A Pilot Study. J Chiropr Med. 2018 Sep;17(3):182-189. doi: 10.1016/j.jcm.2018.03.003. Epub 2018 Aug 26. PMID 30228809
- [Background] Dalal K, Maran VB, Pandey RM, Tripathi M. Determination of efficacy of reflexology in managing patients with diabetic neuropathy: a randomized controlled clinical trial. Evid Based Complement Alternat Med. 2014;2014:843036. doi: 10.1155/2014/843036. Epub 2014 Jan 9. PMID 24527055
- [Background] Wandell PE, Carlsson AC, Gafvels C, Andersson K, Tornkvist L. Measuring possible effect on health-related quality of life by tactile massage or relaxation in patients with type 2 diabetes. Complement Ther Med. 2012 Feb-Apr;20(1-2):8-15. doi: 10.1016/j.ctim.2011.09.007. Epub 2011 Oct 22. PMID 22305243
- [Background] Gok Metin Z, Arikan Donmez A, Izgu N, Ozdemir L, Arslan IE. Aromatherapy Massage for Neuropathic Pain and Quality of Life in Diabetic Patients. J Nurs Scholarsh. 2017 Jul;49(4):379-388. doi: 10.1111/jnu.12300. Epub 2017 Jun 12. PMID 28605119